CLINICAL TRIAL: NCT00961233
Title: Topical Budesonide Treatment for Eosinophilic Esophagitis (EoE): Esophageal Medication Distribution, Treatment Response, and Effect on the Adrenal Axis.
Brief Title: Topical Budesonide Treatment for Eosinophilic Esophagitis (EoE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Evan Dellon, MD, MPH, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRUSESOM0609
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Eosinophilic Esophagitis
Keywords: eosinophilic esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- inhaled/swallowed budesonide (Experimental)
  Interventions: Drug: inhaled/swallowed budesonide
- viscous/swallowed budesonide (Active Comparator)
  Interventions: Drug: viscous/swallowed budesonide

INTERVENTIONS:
Drug: inhaled/swallowed budesonide — medication will be nebulized and then swallowed
  Arms: inhaled/swallowed budesonide
Drug: viscous/swallowed budesonide — viscous suspension of budesonide will be swallowed
  Arms: viscous/swallowed budesonide

SUMMARY:
The purpose of this study is to conduct a clinical trial of two formulations of budesonide (nebulized/swallowed versus viscous/swallowed) in patients with EoE to determine if medication contact time and distribution in the esophagus relates to treatment response. The investigators will also determine if there is systemic absorption of these topical steroids. The investigators hypothesize that tissue and symptom response will correlate with esophageal medication contact time and distribution, and that significant systemic absorption will not be seen.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of eosinophilic esophagitis (per 2007 consensus guidelines)

Exclusion Criteria:

* Age < 18
* Inability to read or understand English
* Pregnant or nursing women
* Previous allergic reactions to steroid medications
* Current use of systemic steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan S Dellon, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Dellon ES, Sheikh A, Speck O, Woodward K, Whitlow AB, Hores JM, Ivanovic M, Chau A, Woosley JT, Madanick RD, Orlando RC, Shaheen NJ. Viscous topical is more effective than nebulized steroid therapy for patients with eosinophilic esophagitis. Gastroenterology. 2012 Aug;143(2):321-4.e1. doi: 10.1053/j.gastro.2012.04.049. Epub 2012 May 3. PMID 22561055

RESULTS

PARTICIPANT FLOW:
Groups:
- Inhaled/Swallowed Budesonide: inhaled/swallowed budesonide - nebulized budesonide 1mg twice daily that is swallowed.
- Viscous/Swallowed Budesonide: viscous/swallowed budesonide - budesonide slurry (created with 5g sucralose) 1 mg twice daily that is swallowed
Period: Overall Study
Arm/Group | Inhaled/Swallowed Budesonide | Viscous/Swallowed Budesonide
Started | 13 | 12
Completed | 11 | 11
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled/Swallowed Budesonide | Viscous/Swallowed Budesonide | Total
Number analyzed (Participants) | 13 | 12 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 34.9 (7.3) | 34.4 (7.5) | 34.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 7 | 15

OUTCOME MEASURES:

1. Secondary Outcome: Adrenal Insufficiency
Description: Adrenal insufficiency as measured by a standard cortisol stimulation test (using 0.25 mg cosyntropin IV and baseline and 60 minute post-injection serum cortisol measurements) after treatment. A rise in serum cortisol concentration after to a peak of ≥18 mcg/dL was considered normal; a smaller rise than this was considered adrenal insufficiency.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Inhaled/Swallowed Budesonide | Viscous/Swallowed Budesonide
Number analyzed (Participants) | 11 | 11
participants | 0 | 0

2. Primary Outcome: Tissue Eosinophil Counts
Description: Level of tissue eosinophil counts (measured in number of eosinophils per high-power microscopy field) on esophageal biopsy after treatment
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: # of eosinophils per high-power field
Groups:
- Inhaled/Swallowed Budesonide: nebulized then swallowed budesonide 1mg twice daily
- Viscous/Swallowed Budesonide: viscous slurry of budesonide and sucralose 1 mg twice daily
Arm/Group | Inhaled/Swallowed Budesonide | Viscous/Swallowed Budesonide
Number analyzed (Participants) | 11 | 11
# of eosinophils per high-power field | 89 (94) | 11 (23)

ADVERSE EVENTS:
Arm/Group | Inhaled/Swallowed Budesonide | Viscous/Swallowed Budesonide
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No